CLINICAL TRIAL: NCT01707186
Title: Pictorial Representation of Illness and Self Measure
Acronym: PRISM
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010930
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2017-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1A: Early phase, requiring change in treatment
- Group 2: Established phase, stable treatment
- Group 2A: Established phase, requiring a change in treatment
- Group 1: Early phase, stable treatment

SUMMARY:
PRISM (Pictorial Representation of Illness and Self Measure) has been developed since the mid-1990s; the task was first developed as a simple measure of how a person was coping with his or her experience of illness. This is an international, multicentre study to evaluate the PRISM tool for the assessment of suffering in rheumatoid arthritis at different stages of the illness and the effect of treatment intervention. There are 5 sites: Berlin, Oxford, Limoges, Montreal and Queensland. The study will recruit 200 patients in total.

In addition to the procedures for the patient's routine clinical visit, the patients will be invited to answer a series of questionnaires and donate 20ml blood sample. Patients will be asked to attend 3 times over 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Written confirmed diagnosed of rheumatoid arthritis

Exclusion Criteria:

* A diagnosis of any of the following:
* Multiple sclerosis
* Motor neurone disease
* Parkinson's disease
* Alzheimer's disease
* Depression or anxiety disorders as identified using the Patient depression screening questions from the patient health questionnaire 9 (PHQ9).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis from hospital clinics
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2012-10-18 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
PRISM/PRISM+ | 30 September 2015
  Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Peter Taylor, FRCP, PhD, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Orthopaedic Centre, Oxford, United Kingdom